CLINICAL TRIAL: NCT03814499
Title: A Multicentre Longitudinal, Observational Natural History Study to Evaluate Disease Progression in Subjects With Usher Syndrome Type 1B (USH1B)
Brief Title: Natural History Study in Subjects With Usher Syndrome
Status: Completed | Type: Observational
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Other Study IDs: TIGEM3-UshTher-NHS
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Usher Syndrome, Type 1B
MeSH Terms: conditions — Usher syndrome, type 1B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Natural History Study in Subjects With Usher Syndrome ((USH1B) is a multi-centre, longitudinal, observational study designed to evaluate disease progression in subjects with USH1B by several vision-related assessments.

DETAILED DESCRIPTION:
Natural History Study in Subjects With Usher Syndrome (USH1B) is being conducted to understand the progression of disease in USH1B patients as measured by visual acuity and visual field testing and a number of other vision-related assessments. Disease progression will be evaluated as change over time in these measures and associations between the endpoints will be examined.

The primary objective of this study is to evaluate the natural progression of disease over time in USHIB patients using visual field testing and best corrected visual acuity.

The secondary objectives of this study are to evaluate the progression of disease over time in USHIB patients through additional assessments:

* Microperimetry (only in selected centres)
* Fundus autofluorescence (FAF)
* Optical Coherence Tomography (OCT)
* Full-field Electroretinogram (ERG),
* Multifocal Electroretinogram,
* Vision-related function and quality of life, as measured by the 25-Item National Eye Institute Visual Function Questionnaire (NEI VFQ-25)

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to adhere to protocol for long-term follow-up as evidenced by written informed consent or parental permission and subject assent.
2. Subjects diagnosed with USH1.
3. Molecular diagnosis of USH1B due to MYO7A mutations (homozygotes or compound heterozygotes).
4. Age eight years old or older at the time of baseline.
5. Visual acuity ≥ 20/640 in at least one eye

Exclusion Criteria:

1. Unable or unwilling to meet requirements of the study.
2. Unable to communicate with suitable verbal/auditory and/or tactile sign language (in the opinion of the investigator)
3. Participation in a clinical study with an investigational drug in the past six months.
4. Pre-existing eye conditions that would interfere with the interpretation of study endpoints (for example, glaucoma, corneal or significant lenticular opacities, cystoid macular oedema, macular hole).
5. Complicating systemic diseases in which the disease itself, or the treatment for the disease, can alter ocular function. Examples are malignancies whose treatment could affect central nervous system function (for example, radiation treatment of the orbit; leukemia with CNS/optic nerve involvement). Also excluded would be subjects with immuno- compromising diseases, as there could be susceptibility to opportunistic infection [such as cytomegalovirus (CMV) retinitis].
6. Subjects with diabetes or sickle cell disease would be excluded if they had any manifestation of advanced retinopathy (e.g. macular edema or proliferative changes).
7. Prior ocular surgery within three months.
8. Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study and, in the opinion of the investigator, makes the potential subject unsuitable for the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects affected by Usher Syndrome 1B disease fulfilled eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FRANCESCA SIMONELLI, Principal Investigator — Eye Clinic of the University of Campania Luigi Vanvitelli, Naples, Italy; Ingeborgh van den Born, Principal Investigator — Stichting Oogziekenhuis Rotterdam, Rotterdam, The Netherland.; Carmen Ayuso, Principal Investigator — Instituto de Investigacion Sanitaria de la Fundacion Jimenez Diaz, Madrid, Spain
Locations (3):
- Eye Clinic of the University of Campania Luigi Vanvitelli, Naples, Italy
- Stichting Oogziekenhuis Rotterdam, Rotterdam, Netherlands
- Instituto de Investigacion Sanitaria de la Fundacion Jimenez Diaz, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 53 subjects meeting the inclusion/exclusion criteria were enrolled in the 18-month recruitment period.
Groups:
- Group of Subjects With Usher Syndrome Type 1B: In this study, there is 1 group of subjects with Usher Syndrome type 1B enrolled, over the 18-month recruitment period, to evaluate disease progression by several vision-related assessments.
  Subjects will be assessed using the following schedule:
  * Baseline visit
  * 1 year follow-up visit
  * 2 year follow-up visit
Period: Overall Study
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Started | 53 (53 patients were enrolled at Baseline visit.)
Completed | 50 (1. patient lost to follow up at 1 year visit; 2. patients lost to follow up at 2 years visit.)
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: A total of 61 patients (32 screened by Unicamp, 20 by IIS-FJD and 9 by REH) with clinical diagnosis of USH1 were screened for inclusion in the study. 8 of these were excluded according to exclusion/inclusion criteria.
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants] — Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Participants
    <=18 years | 11
    Between 18 and 65 years | 39
    >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  years | 33.6 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Participants
    Female | 23
    Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 53
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion/exclusion criteria.
  participants
    Netherlands | 8
    Italy | 29
    Spain | 16
BCVA - better seeing eyes [Mean (Standard Deviation); unit: ETDRS Score] — Best Corrected Visual acuity in the better-seeing eyes. The ETDRS score (minimum value 0 and maximum value 100, with 0 representing the worst, and 100 the best visual functioning) is calculated as the total number of letters correctly read at 4m from the chart plus 30 (if 20 or more letters can be read at 4m). If fewer than 20 letters can be read at 4m, the patient's position is adjusted to 1m in front of the chart. Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion/exclusion criteria.
  ETDRS Score | 66.4 (17.9)
III4e Area - better seeing eyes [Mean (Standard Deviation); unit: Degree Squared] — Visual field area using III4e stimulus size in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Degree Squared | 3365.8 (4142.1)
V4e Area - better seeing eyes [Mean (Standard Deviation); unit: Degree squared] — Visual field area using V4e stimulus size in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Degree squared | 5605.2 (5290.2)
MS - better seeing eyes [Mean (Standard Deviation); unit: Decibels] — Macular sensitivity, assessed by microperimetry, in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Decibels | 9.7 (9.9)
CMT - better seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Central Macular Thickness, evaluated with Optical Coherence tomography, in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 259.6 (63)
EZ Band Horizontal - better seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 2807.5 (2374.6)
EZ Band Vertical - better seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (vertical scan), in the better-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 2436.1 (2286.4)
BCVA - worse seeing eyes [Mean (Standard Deviation); unit: ETDRS score] — Best Corrected Visual acuity in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  ETDRS score | 59.5 (21.7)
III4e Area - worse seeing eyes [Mean (Standard Deviation); unit: Degree squared] — Visual field area using III4e stimulus size in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Degree squared | 4176.4 (4400.3)
V4e Area - worse seeing eyes [Mean (Standard Deviation); unit: Degree squared] — Visual field area using V4e stimulus size in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Degree squared | 5613.22 (5127.2)
MS - worse seeing eyes [Mean (Standard Deviation); unit: Decibels] — Macular sensitivity, assessed by microperimetry, in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Decibels | 9 (10.2)
CMT - worse seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Central Macular Thickness, evaluated with Optical Coherence tomography, in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 250.7 (63.3)
EZ Hor. - worse seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 2615.5 (2370.4)
EZ Vert. - worse seeing eyes [Mean (Standard Deviation); unit: Micrometers] — Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (vertical scan), in the worse-seeing eyes Population: As mentioned before, 61 patients were screened, but 53 patients were considered for analyses because 8 patients did not meet the inclusion criteria.
  Micrometers | 2332.4 (666.5)

OUTCOME MEASURES:

1. Primary Outcome: BCVA - Better Seeing Eyes
Description: Change (from Baseline) in Best Corrected Visual acuity (BCVA) in the better-seeing eyes.
  BCVA in the better seeing eyes was assessed using the ETRS score (minimum value 0 and maximum value 100, with 0 representing the worst, and 100 the best visual functioning).
  The results are reported as the change in ETDRS score collected at the 1 year follow-up visit compared with the score at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visit
Measure: Mean (Standard Deviation); unit: ETDRS score
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
ETDRS score | -2.26 (3.838)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p < 0.01, Regression, Linear; Coefficient = -2.3

2. Primary Outcome: BCVA - Better Seeing Eyes
Description: Change (from Baseline) in Best Corrected Visual acuity (BCVA) in the better-seeing eyes.
  BCVA in the better seeing eyes was assessed using the ETRS score (minimum value 0 and maximum value 100, with 0 representing the worst, and 100 the best visual functioning).
  The results are reported as the change in ETDRS score collected at the 2 year follow-up visit compared with the score at the baseline visit.
Time Frame: 2 year follow up visit
Population: patients undergoing two-year follow-up visit
Measure: Mean (Standard Deviation); unit: ETDRS score
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
ETDRS score | -1.468 (4.999)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p < 0.01, Regression, Linear; Coefficient = -3.8

3. Primary Outcome: III4e Area - Better Seeing Eyes
Description: Change (from Baseline) in visual field area using III4e stimulus size in the better seeing eyes.
  Visual field area using III4e stimulus size in the better seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
degree squared | 561.966 (2043.612)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.3269, Regression, Linear; Coefficient = 369.9

4. Primary Outcome: III4e Area - Better Seeing Eyes
Description: Change (from Baseline) in visual field area using III4e stimulus size in the better seeing eyes.
  Visual field area using III4e stimulus size in the better seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 year follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
degree squared | 70.286 (1451.128)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.4265, Regression, Linear; Coefficient = 365.4

5. Primary Outcome: V4e Area - Better Seeing Eyes
Description: Change (from Baseline) in visual field area using V4e stimulus size in the better seeing eyes.
  Visual field area using V4e stimulus size in the better seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
degree squared | 273.309 (2432.785)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.4782, Regression, Linear; Coefficient = 264.3

6. Primary Outcome: V4e Area - Better Seeing Eyes
Description: Change (from Baseline) in visual field area using V4e stimulus size in the better seeing eyes.
  Visual field area using V4e stimulus size in the better seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 year follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
degree squared | 700.245 (3942.6)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.2716, Regression, Linear; Coefficient = 730.2

7. Primary Outcome: BCVA - Worse Seeing Eyes
Description: Change (from Baseline) in Best Corrected Visual acuity (BCVA) in the worse seeing eyes.
  BCVA in the worse seeing eyes was assessed using the ETRS score (minimum value 0 and maximum value 100, with 0 representing the worst, and 100 the best visual functioning).
  The results are reported as the change in the ETDRS score collected at the 1 year follow-up visit compared with the score at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: ETDRS score
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
ETDRS score | -0.625 (5.35)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.4178, Regression, Linear; Coefficient = -0.6

8. Primary Outcome: BCVA - Worse Seeing Eyes
Description: Change (from Baseline) in Best Corrected Visual acuity in the worse seeing eyes.
  Best corrected visual acuity in the worse seeing eyes was assessed using the ETRS score (minimum value 0 and maximum value 100, with 0 representing the worst, and 100 the best visual functioning).
  The results are reported as the change in the ETDRS score collected at the 2 year follow-up visit compared with the score at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: ETDRS score
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
ETDRS score | -0.909 (7.041)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.2677, Regression, Linear; Coefficient = -1.5

9. Primary Outcome: III4e Area - Worse Seeing Eyes
Description: Change (from Baseline) in visual field area using III4e stimulus size in the worse-seeing eyes.
  Visual field area using III4e stimulus size in the worse-seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
degree squared | -445.569 (2920.491)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.3364, Regression, Linear; Coefficient = -467

10. Primary Outcome: III4e Area - Worse Seeing Eyes
Description: Change (from Baseline) in visual field area using III4e stimulus size in the worse-seeing eyes.
  Visual field area using III4e stimulus size in the worse-seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
degree squared | -407.928 (3209.147)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.1124, Regression, Linear; Coefficient = -908

11. Primary Outcome: V4e Area - Worse Seeing Eyes
Description: Change (from Baseline) in visual field area using V4e stimulus size in the worse-seeing eyes.
  Visual field area using V4e stimulus size in the worse-seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
degree squared | 391.212 (2726.331)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.2649, Regression, Linear; Coefficient = 479.2

12. Primary Outcome: V4e Area - Worse Seeing Eyes
Description: Change (from Baseline) in visual field area using V4e stimulus size in the worse-seeing eyes.
  Visual field area using V4e stimulus size in the worse-seeing eyes is expressed in degree squared (minimum value 0, maximum value 20000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: degree squared
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
degree squared | 610.017 (5658.524)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.216, Regression, Linear; Coefficient = 1114.3

13. Secondary Outcome: MS - Better Seeing Eyes
Description: Change (from Baseline) in macular sensitivity, assessed by microperimetry, in the better-seeing eyes.
  Macular sensitivity, assessed by microperimetry is expressed in decibels (minimum value 0, maximum value 30).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
decibels | 0.137 (2.89)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.9032, Regression, Linear; Coefficient = 0.1

14. Secondary Outcome: MS - Better Seeing Eyes
Description: Change (from Baseline) in macular sensitivity, assessed by microperimetry, in the better-seeing eyes.
  Macular sensitivity, assessed by microperimetry is expressed in decibels (minimum value 0, maximum value 30).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
decibels | -0.315 (7.174)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.7889, Regression, Linear; Coefficient = -0.4

15. Secondary Outcome: CMT - Better Seeing Eyes
Description: Change (from Baseline) in Central Macular Thickness (CMT), evaluated with Optical Coherence tomography, in the better-seeing eyes.
  CMT was reported in micrometers (minimum value 0, maximum value 1000). The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | 7 (21.532)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.0242, Regression, Linear; Coefficient = 7

16. Secondary Outcome: CMT - Better Seeing Eyes
Description: Change (from Baseline) in Central Macular Thickness (CMT), evaluated with Optical Coherence tomography, in the better-seeing eyes.
  CMT was reported in micrometers (minimum value 0, maximum value 1000). The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | -5.667 (18.877)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.5092, Regression, Linear; Coefficient = 1.5

17. Secondary Outcome: EZ Band Horizontal - Better Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the better-seeing eyes.
  EZ Band Horizontal is reported in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | -42.795 (324.893)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.3634, Regression, Linear; Coefficient = -47.1

18. Secondary Outcome: EZ Band Horizontal - Better Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the better-seeing eyes.
  EZ Band Horizontal is reported in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | -160.556 (628.761)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.0677, Regression, Linear; Coefficient = -204.7

19. Secondary Outcome: EZ Band Vertical - Better Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (Vertical scan), in the better-seeing eyes.
  EZ Band Vertical is reported in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | -289.75 (1107.784)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.156, Regression, Linear; Coefficient = -235.8

20. Secondary Outcome: EZ Band Vertical - Better Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (Vertical scan), in the better-seeing eyes.
  EZ Band Vertical is reported in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | 190.553 (1276.729)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.3148, Regression, Linear; Coefficient = -102

21. Secondary Outcome: MS - Worse Seeing Eyes
Description: Change (from Baseline) in macular sensitivity, assessed by microperimetry, in the worse-seeing eyes.
  Macular sensitivity, assessed by microperimetry is expressed in decibels (minimum value 0, maximum value 30).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
decibels | -0.056 (3.279)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.9349, Regression, Linear; Coefficient = -0.1

22. Secondary Outcome: MS - Worse Seeing Eyes
Description: Change (from Baseline) in macular sensitivity, assessed by microperimetry, in the worse-seeing eyes.
  Macular sensitivity, assessed by microperimetry is expressed in decibels (minimum value 0, maximum value 30).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: decibels
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
decibels | -0.758 (7.062)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.7196, Regression, Linear; Coefficient = -0.6

23. Secondary Outcome: CMT - Worse Seeing Eyes
Description: Change (from Baseline) in Central Macular Thickness (CMT), evaluated with Optical Coherence tomography, in the worse-seeing eyes.
  CMT is expressed in micrometers (minimum value 0, maximum value 1000). The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | 4.786 (15.682)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.0542, Regression, Linear; Coefficient = 4.7

24. Secondary Outcome: CMT - Worse Seeing Eyes
Description: Change (from Baseline) in Central Macular Thickness, evaluated with Optical Coherence tomography, in the worse-seeing eyes.
  CMT is expressed in micrometers (minimum value 0, maximum value 1000). The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | -2.026 (22.358)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.4224, Regression, Linear; Coefficient = 2.6

25. Secondary Outcome: EZ Band Horizontal - Worse Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the worse-seeing eyes.
  EZ Band Horizontal is expressed in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | -122.763 (486.734)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.1247, Regression, Linear; Coeffiient = -118.9

26. Secondary Outcome: EZ Band Horizontal - Worse Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (horizontal scan), in the worse-seeing eyes.
  EZ Band Horizontal is expressed in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | -21.658 (237.373)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.1461, Regression, Linear; Coefficient = -135.2

27. Secondary Outcome: EZ Band Vertical - Worse Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (Vertical scan), in the worse-seeing eyes.
  EZ Band Vertical is expressed in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 1 year follow-up visit compared with the values at the baseline visit.
Time Frame: 1 year follow up visit
Population: patients undergoing one-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 52
micrometers | -149.051 (528.203)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.0699, Regression, Linear; Coefficient = -154.2

28. Secondary Outcome: EZ Band Vertical - Worse Seeing Eyes
Description: Change (from Baseline) in Ellipsoid Zone Band Width, evaluated with Optical Coherence tomography (Vertical scan), in the worse-seeing eyes.
  EZ Band Vertical is expressed in micrometers (minimum value 0, maximum value 4000).
  The results are reported as the change in the values collected at the 2 year follow-up visit compared with the values at the baseline visit.
Time Frame: 2 years follow up visit
Population: patients undergoing two-year follow-up visits
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
Number analyzed (Participants) | 50
micrometers | -15.861 (236.02)
Statistical Analysis 1: Comparison: Group of Subjects With Usher Syndrome Type 1B; Test type: Other; p = 0.0901, Regression, Linear; Coefficient = -164.6

ADVERSE EVENTS:
Time Frame: 1 year, 2 years
Groups:
- Group of Subjects With Usher Syndrome Type 1B: In this study, there is 1 group of subjects with Usher Syndrome type 1B enrolled, over the 18-month recruitment period, to evaluate disease progression by several vision-related assessments.
  Subjects will be assessed using the following schedule:
  * 1 year follow-up visit
  * 2 year follow-up visit
Arm/Group | Group of Subjects With Usher Syndrome Type 1B
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03814499/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT03814499/ICF_001.pdf